CLINICAL TRIAL: NCT00762801
Title: Studies on the Expression and Functions of RLIP76 in Blood Samples of Healthy Human Subjects
Status: Withdrawn | Type: Observational
Why Stopped: Principal Investigator left institution.
Sponsor: University of North Texas Health Science Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-32
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: RLIP76; Cancer; apoptosis
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
RLIP76 (Ral binding protein1) is a 76 kDa splice variant protein encoded by the human gene (RALBP1, 18p11.22). It is a multifunctional modular protein found ubiquitously from Drosophila to humans, in cells ranging from red blood cells to endothelial cells of the brain. Its expression more predominant in breast, heart, liver and less so in colon and brain parenchyma.

DETAILED DESCRIPTION:
RLIP76 is shown to be over expressed in a variety of cancer cells. However, no study has yet been done on its expression on normal cells. The studies proposed in this project will study the expression of RLIP76 in blood cells of healthy human subjects in the population of North Texas region.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as defined by lack of serious health conditions or diseases

Exclusion Criteria:

* Children, pregnant women, prisoners, persons with any medical condition that precludes phlebotomy and persons unwilling or unable to provide consent will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 healthy volunteers
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Expression of RLIP76 in red blood cells and white blood cells of 100 healthy human subjects. | 3 years

SECONDARY OUTCOMES:
To investigate the RLIP76 mediated transport of glutathione conjugates and chemotherapeutic drugs. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Awasthi, MD, Principal Investigator — University of North Texas Health Science Center
Locations (1):
- University of North Texas Health Science Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singhal SS, Yadav S, Singhal J, Zajac E, Awasthi YC, Awasthi S. Depletion of RLIP76 sensitizes lung cancer cells to doxorubicin. Biochem Pharmacol. 2005 Aug 1;70(3):481-8. doi: 10.1016/j.bcp.2005.05.005. PMID 15950949
- [Background] Cheng JZ, Sharma R, Yang Y, Singhal SS, Sharma A, Saini MK, Singh SV, Zimniak P, Awasthi S, Awasthi YC. Accelerated metabolism and exclusion of 4-hydroxynonenal through induction of RLIP76 and hGST5.8 is an early adaptive response of cells to heat and oxidative stress. J Biol Chem. 2001 Nov 2;276(44):41213-23. doi: 10.1074/jbc.M106838200. Epub 2001 Aug 24. PMID 11522795
- [Background] Awasthi S, Singhal SS, Srivastava SK, Zimniak P, Bajpai KK, Saxena M, Sharma R, Ziller SA 3rd, Frenkel EP, Singh SV, et al. Adenosine triphosphate-dependent transport of doxorubicin, daunomycin, and vinblastine in human tissues by a mechanism distinct from the P-glycoprotein. J Clin Invest. 1994 Mar;93(3):958-65. doi: 10.1172/JCI117102. PMID 7907606
- [Background] Awasthi S, Singhal SS, Pikula S, Piper JT, Srivastava SK, Torman RT, Bandorowicz-Pikula J, Lin JT, Singh SV, Zimniak P, Awasthi YC. ATP-Dependent human erythrocyte glutathione-conjugate transporter. II. Functional reconstitution of transport activity. Biochemistry. 1998 Apr 14;37(15):5239-48. doi: 10.1021/bi972131r. PMID 9548755
- [Background] Zou W, Borvak J, Marches F, Wei S, Galanaud P, Emilie D, Curiel TJ. Macrophage-derived dendritic cells have strong Th1-polarizing potential mediated by beta-chemokines rather than IL-12. J Immunol. 2000 Oct 15;165(8):4388-96. doi: 10.4049/jimmunol.165.8.4388. PMID 11035076
- [Result] McIlwain CC, Townsend DM, Tew KD. Glutathione S-transferase polymorphisms: cancer incidence and therapy. Oncogene. 2006 Mar 13;25(11):1639-48. doi: 10.1038/sj.onc.1209373. PMID 16550164
- [Result] Jullien-Flores V, Mahe Y, Mirey G, Leprince C, Meunier-Bisceuil B, Sorkin A, Camonis JH. RLIP76, an effector of the GTPase Ral, interacts with the AP2 complex: involvement of the Ral pathway in receptor endocytosis. J Cell Sci. 2000 Aug;113 ( Pt 16):2837-44. doi: 10.1242/jcs.113.16.2837. PMID 10910768
- [Result] Awasthi S, Cheng J, Singhal SS, Saini MK, Pandya U, Pikula S, Bandorowicz-Pikula J, Singh SV, Zimniak P, Awasthi YC. Novel function of human RLIP76: ATP-dependent transport of glutathione conjugates and doxorubicin. Biochemistry. 2000 Aug 8;39(31):9327-34. doi: 10.1021/bi992964c. PMID 10924126
- [Result] Awasthi S, Sharma R, Singhal SS, Zimniak P, Awasthi YC. RLIP76, a novel transporter catalyzing ATP-dependent efflux of xenobiotics. Drug Metab Dispos. 2002 Dec;30(12):1300-10. doi: 10.1124/dmd.30.12.1300. PMID 12433796
- [Result] Awasthi S, Singhal SS, Yadav S, Singhal J, Drake K, Nadkar A, Zajac E, Wickramarachchi D, Rowe N, Yacoub A, Boor P, Dwivedi S, Dent P, Jarman WE, John B, Awasthi YC. RLIP76 is a major determinant of radiation sensitivity. Cancer Res. 2005 Jul 15;65(14):6022-8. doi: 10.1158/0008-5472.CAN-05-0968. PMID 16024601
- [Result] Yadav S, Zajac E, Singhal SS, Awasthi S. Linking stress-signaling, glutathione metabolism, signaling pathways and xenobiotic transporters. Cancer Metastasis Rev. 2007 Mar;26(1):59-69. doi: 10.1007/s10555-007-9043-5. PMID 17260165
- [Result] Jullien-Flores V, Dorseuil O, Romero F, Letourneur F, Saragosti S, Berger R, Tavitian A, Gacon G, Camonis JH. Bridging Ral GTPase to Rho pathways. RLIP76, a Ral effector with CDC42/Rac GTPase-activating protein activity. J Biol Chem. 1995 Sep 22;270(38):22473-7. doi: 10.1074/jbc.270.38.22473. PMID 7673236
- [Result] Shurin GV, Tourkova IL, Chatta GS, Schmidt G, Wei S, Djeu JY, Shurin MR. Small rho GTPases regulate antigen presentation in dendritic cells. J Immunol. 2005 Mar 15;174(6):3394-400. doi: 10.4049/jimmunol.174.6.3394. PMID 15749872
- [Result] DODGE JT, MITCHELL C, HANAHAN DJ. The preparation and chemical characteristics of hemoglobin-free ghosts of human erythrocytes. Arch Biochem Biophys. 1963 Jan;100:119-30. doi: 10.1016/0003-9861(63)90042-0. No abstract available. PMID 14028302
- [Result] Stuckler D, Singhal J, Singhal SS, Yadav S, Awasthi YC, Awasthi S. RLIP76 transports vinorelbine and mediates drug resistance in non-small cell lung cancer. Cancer Res. 2005 Feb 1;65(3):991-8. PMID 15705900
- [Result] Singhal SS, Wickramarachchi D, Singhal J, Yadav S, Awasthi YC, Awasthi S. Determinants of differential doxorubicin sensitivity between SCLC and NSCLC. FEBS Lett. 2006 Apr 17;580(9):2258-64. doi: 10.1016/j.febslet.2006.03.038. Epub 2006 Mar 24. PMID 16579994
- [Result] Boyum A, Lovhaug D, Tresland L, Nordlie EM. Separation of leucocytes: improved cell purity by fine adjustments of gradient medium density and osmolality. Scand J Immunol. 1991 Dec;34(6):697-712. doi: 10.1111/j.1365-3083.1991.tb01594.x. PMID 1749920
- [Result] Bradford MM. A rapid and sensitive method for the quantitation of microgram quantities of protein utilizing the principle of protein-dye binding. Anal Biochem. 1976 May 7;72:248-54. doi: 10.1016/0003-2697(76)90527-3. No abstract available. PMID 942051
- [Result] Laemmli UK. Cleavage of structural proteins during the assembly of the head of bacteriophage T4. Nature. 1970 Aug 15;227(5259):680-5. doi: 10.1038/227680a0. No abstract available. PMID 5432063
- [Result] Towbin H, Staehelin T, Gordon J. Electrophoretic transfer of proteins from polyacrylamide gels to nitrocellulose sheets: procedure and some applications. Proc Natl Acad Sci U S A. 1979 Sep;76(9):4350-4. doi: 10.1073/pnas.76.9.4350. PMID 388439
- [Result] Steck TL, Kant JA. Preparation of impermeable ghosts and inside-out vesicles from human erythrocyte membranes. Methods Enzymol. 1974;31:172-80. doi: 10.1016/0076-6879(74)31019-1. No abstract available. PMID 4370662